CLINICAL TRIAL: NCT02799823
Title: Transfemoral Replacement of Aortic Valve With HLT MeriDIAN Valve Early Feasibility Trial
Acronym: RADIANT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: HLT Business Decision
Sponsor: HLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLT1501
Record Dates: First submitted 2016-06-03; First posted 2016-06-15 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Aortic Valve Stenosis
Keywords: aortic stenosis; transcatheter aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- HLT Transcatheter Aortic Valve System (Experimental): Transcatheter aortic valve replacement with HLT Transcatheter Aortic Valve System
  Interventions: Device: HLT Transcatheter Aortic Valve System

INTERVENTIONS:
Device: HLT Transcatheter Aortic Valve System — Transcatheter aortic valve replacement with HLT Transcatheter Aortic Valve System

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the HLT System in patients with severe aortic stenosis who present at High Risk for aortic valve replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 70 years of age or older
2. Echocardiographic or hemodynamic based evidence of calcific (senile) aortic stenosis with one of the following: aortic valve EOA <1.0 cm2 or 0.6 cm2/m2, mean aortic valve gradient >40 mmHg or peak aortic valve velocity >4 m/sec
3. Symptoms due to aortic stenosis resulting in one of the following:

   1. New York Heart Association (NYHA) Functional Classification of II or greater
   2. Presence of angina
   3. Presence of syncope
4. Documented aortic valve annular diameter ≥ 21 and ≤ 24 mm (associated perimeter range is 66.0 - 75.4 mm or associated area range of 346 - 452 mm2) measured by the multislice computed tomography (MSCT) Core Lab assessment of pre-procedure imaging.
5. Documented heart team agreement of high risk for surgical aortic valve replacement (SAVR) due to frailty or comorbidities such as:

   * Society of Thoracic Surgeons (STS) score of ≥8%
   * Frailty as indicated by one of the following:

     * Five meter walk test > 6 seconds
     * Katz activities of daily living (ADL) score of 3/6 or less
     * Body Mass Index < 20 kg/m2
     * Wheelchair bound, unable to live independently
   * Childs Class A or B liver disease
   * Severe lung disease (need for supplemental oxygen, forced expiratory volume at one second (FEV1) < 50% of predicted, diffusing capacity of the lungs for carbon monoxide (DLCO) < 60%, or other evidence of severe pulmonary dysfunction
   * Previous coronary artery bypass graft(s) at risk for re-operation
   * Serum albumin < 3.5 g/dL
   * Other evidence that subject is at high risk for surgical valve replacement by one of the following:

     * Hostile chest
     * Porcelain aorta
     * Severe pulmonary hypertension (> 60 mmHg)
     * Prior chest radiation therapy
     * Neuromuscular disease that creates risk for mechanical ventilation or rehabilitation after surgical aortic valve replacement
     * Orthopedic disease that creates risk for rehabilitation after surgical aortic valve replacement
6. Geographically available, willing to comply with follow up and able to provide written informed consent

Exclusion Criteria:

1. Congenital unicuspid or bicuspid aortic valve, or noncalcified aortic valve; or valve eccentricity (calcific or otherwise) which could compromise procedural success.
2. Patients with a coronary height of < 10mm, or otherwise determined to be high risk for coronary obstruction
3. Patients with low flow/low gradient aortic stenosis
4. Patients with significant annular or left ventricular outflow tract (LVOT) calcification that could compromise procedural success
5. Pre-existing prosthetic heart valve in any position
6. Severe aortic, mitral or tricuspid valve regurgitation
7. Moderate to severe mitral stenosis
8. Myocardial infarction within the past 30 days*
9. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
10. Left Ventricular Ejection Fraction (LVEF) < 30%
11. Severe pulmonary hypertension with pulmonary systolic pressure greater than two- thirds of systemic pressure
12. Hemodynamic instability requiring inotropic drug therapy within the past 14 days
13. Untreated clinically significant coronary artery disease requiring revascularization
14. Presence of significant aortic disease such as atheroma, thrombus, or aneurysm which precludes safe implant delivery
15. Blood dyscrasias defined as leukopenia (White blood cell count < 1,000 cell/mm3), anemia (hemoglobin < 9.0 g/dL), thrombocytopenia (platelet count < 50,000 cells/mm3), history of bleeding diathesis or coagulopathy
16. Patient ineligible for or refuses blood transfusions
17. Unfavorable peripheral vascular anatomy or disease (e.g. severe obstructive calcification, severe tortuosity) that would preclude passage of 18 French (18F) catheters from the femoral arterial access to the aorta as evidenced by peripheral MSCT
18. Active peptic ulcer or gastrointestinal bleeding within the past 90 days, that would not allow treatment with the protocol antiplatelet regimen post implant *
19. Symptoms of carotid or vertebral artery disease (e.g. stroke or transient ischemic attack) within past 6 months, or treatment of carotid stenosis within past two months*
20. Renal disease as demonstrated by a serum creatinine > 2.5 mg/dL or end stage renal disease
21. Active infection (including endocarditis) requiring ongoing treatment
22. Need for emergent surgery or intervention other than the investigational procedure
23. Any therapeutic invasive cardiac procedure performed or planned to perform within 30 days of the index procedure, except for percutaneous coronary intervention (PCI) which is performed within 7 days prior to the index procedure*
24. Hypersensitivity or contraindication to procedural medication and device materials (e.g. titanium, nickel, pork) which cannot be adequately premedicated
25. Life expectancy < 1 year due to non-cardiac co-morbid conditions
26. Currently participating in any investigational drug or device studies that may confound the results of this study
27. History of any cognitive or mental health status that would interfere with study participation
28. Following surgical consultation, patient is deemed inoperable in the event that surgical intervention is required after Meridian valve implantation
29. Patients with a history of hypertrophic cardiomyopathy
30. Aortic root angle ≥ 70˚ as determined by the MSCT Core Lab assessment of pre- procedure imaging
31. Unfavorable left ventricular anatomy (e.g., size or shape) as evidenced by pre- procedure imaging * At the time of procedure, if a subject's medical status has changed since enrollment, the subject shall be re-evaluated for eligibility

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: Mortality at 30 days | 30 days
  The primary safety endpoint is all-cause mortality at 30 days.

SECONDARY OUTCOMES:
Secondary Performance Endpoint 1: Procedural Device Performance | 1 day
  The secondary performance endpoint is Device Success defined as:
  * Absence of procedural mortality AND
  * Correct positioning of a single Valve into the proper anatomical location AND
  * Intended performance of the Valve (no severe prosthesis-patient mismatch and clinically acceptable gradient) AND no moderate or severe aortic valve regurgitation)
Secondary Performance Endpoint 2: Post-procedural Valve Performance | pre-discharge, 1, 6, 12, 24, 36, 48 and 60 months
  The Valve performance will be evaluated by the following parameters with echocardiograms obtained at pre-discharge, 1, 6, 12, 24, 36, 48 and 60 months:
  * Aortic valve effective orifice area (EOA)
  * Severity of aortic valve regurgitation (AR)
  * Aortic valve gradient
Secondary Safety Endpoint 3: Adverse Events | Throughout the 5 year follow up period
  All adverse events will be assessed throughout the 5 year follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Williams, MD, Principal Investigator — NYU Langone Medical Center; Dean Kereiakes, MD, Principal Investigator — The Christ Hospital
Locations (5):
- United States (5):
  - MedStar Health, Washington D.C., District of Columbia
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - NYU Langone Medical Center, New York, New York
  - The Lindner Center for Research and Education at the Christ Hospital, Cincinnati, Ohio
  - Baylor Scott & White The Heart Hospital Plano, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodes-Cabau J, Williams MR, Wijeysundera HC, Kereiakes DJ, Paradis JM, Staniloae C, Saric M, Radhakrishnan S, Wilson RF, Kubo SH. Transcatheter Aortic Valve Replacement With the HLT Meridian Valve. Circ Cardiovasc Interv. 2019 Aug;12(8):e008053. doi: 10.1161/CIRCINTERVENTIONS.119.008053. Epub 2019 Jul 31. PMID 31362540